CLINICAL TRIAL: NCT01375647
Title: Exploration of the Biologic Basis for Underperformance of Oral Polio and Rotavirus Vaccines in Bangladesh
Acronym: PROVIDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Virginia (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Washington University School of Medicine (Other); Stanford University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Beth Kirkpatrick, M.D., University of Vermont
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: PROVIDE
Record Dates: First submitted 2011-06-03; First posted 2011-06-17 (Estimated); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Rotavirus Diarrhea; Vaccine Virus Shedding; Tropical Enteropathy
Keywords: Oral Vaccines; Vaccine Responsiveness; Tropical Enteropathy
MeSH Terms: conditions — Sprue, Tropical | interventions — Poliovirus Vaccine, Inactivated; RIX4414 vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rotarix + No IPV (inactivated polio vaccine) (Experimental): Oral Rotarix vaccine at 10 and 17 weeks of age and oral polio vaccine series
  Interventions: Biological: Rotarix
- Rotarix + IPV (inactivated polio vaccine) (Experimental): Oral Rotarix vaccine at 10 and 17 weeks of age plus IPV (inactivated polio vaccine) boost in place of oral polio vaccine dose at 39 weeks
  Interventions: Biological: IPV (inactivated polio vaccine); Biological: Rotarix
- No Rotarix + No IPV (inactivated polio vaccine) (No Intervention): No Rotarix and oral polio vaccine series only
- No Rotarix + IPV (inactivated polio vaccine) (Experimental): No Rotarix vaccine and IPV (inactivated polio vaccine) boost in place of oral polio vaccine dose at 39 weeks
  Interventions: Biological: IPV (inactivated polio vaccine)

INTERVENTIONS:
Biological: IPV (inactivated polio vaccine) — Administered per protocol
  Arms: No Rotarix + IPV (inactivated polio vaccine); Rotarix + IPV (inactivated polio vaccine)
Biological: Rotarix — Administered per protocol
  Arms: Rotarix + IPV (inactivated polio vaccine); Rotarix + No IPV (inactivated polio vaccine)

SUMMARY:
Oral polio and rotavirus vaccines are significantly less effective in children living in the developing world. Tropical enteropathy, which is associated with intestinal inflammation, decreased absorption and increased permeability, may contribute substantially to oral vaccine failure in developing country settings. Other possible causes of oral vaccine underperformance include malnutrition, interference with maternal or breastmilk antibodies, changes in gut microbiota, and genetic susceptibility.

Primary Objective: to determine whether tropical enteropathy impairs the efficacy of oral polio and rotavirus vaccines in children in Bangladesh.

Secondary Objectives: 1) to determine the impact of an IPV (inactivated polio vaccine) boost on the efficacy of OPV (oral polio vaccine) and 2) to determine the efficacy of Rotarix oral rotavirus vaccine to prevent rotavirus diarrhea

The polio and rotavirus randomized clinical trials are embedded as secondary objectives within the exploratory study of tropical enteropathy. The primary and secondary outcome measures are relevant to the randomized clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Mother willing to sign informed consent form.
2. Healthy infant aged 0 to 7 days old.
3. No obvious congenital abnormalities or birth defects.
4. No abnormal (frequency and consistency) stools since birth.
5. Stable household with no plans to leave the area for the next one year.

Exclusion Criteria:

1. Parents are not willing to have child vaccinated at the field clinic.
2. Parents are not willing to have child's blood drawn.
3. Parents are planning to enroll child into another clinical study during the time period of this trial.
4. Mother not willing to have blood drawn and breast milk extracted.
5. Parents not willing to have field research assistant in home two times per week.
6. History of seizures or other apparent neurologic disorders.
7. Infant received any vaccines before start of study, except Bacillus Calmette-Guerin (BCG).
8. Infant has any sibling currently or previously enrolled in this study, including a twin.

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 700 (Actual)
Dates: Start 2011-05; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Kirkpatrick, M.D., Principal Investigator — University of Vermont; William Petri, M.D., Ph.D., Principal Investigator — University of Virginia School of Medicine; Rashidul Haque, M.D., Ph.D., Principal Investigator — International Center for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

REFERENCES:
- [Background] Kirkpatrick BD, Colgate ER, Mychaleckyj JC, Haque R, Dickson DM, Carmolli MP, Nayak U, Taniuchi M, Naylor C, Qadri F, Ma JZ, Alam M, Walsh MC, Diehl SA; PROVIDE Study Teams; Petri WA Jr. The "Performance of Rotavirus and Oral Polio Vaccines in Developing Countries" (PROVIDE) study: description of methods of an interventional study designed to explore complex biologic problems. Am J Trop Med Hyg. 2015 Apr;92(4):744-51. doi: 10.4269/ajtmh.14-0518. Epub 2015 Feb 23. PMID 25711607
- [Result] Colgate ER, Haque R, Dickson DM, Carmolli MP, Mychaleckyj JC, Nayak U, Qadri F, Alam M, Walsh MC, Diehl SA, Zaman K, Petri WA, Kirkpatrick BD. Delayed Dosing of Oral Rotavirus Vaccine Demonstrates Decreased Risk of Rotavirus Gastroenteritis Associated With Serum Zinc: A Randomized Controlled Trial. Clin Infect Dis. 2016 Sep 1;63(5):634-41. doi: 10.1093/cid/ciw346. Epub 2016 May 23. PMID 27217217
- [Result] Mychaleckyj JC, Haque R, Carmolli M, Zhang D, Colgate ER, Nayak U, Taniuchi M, Dickson D, Weldon WC, Oberste MS, Zaman K, Houpt ER, Alam M, Kirkpatrick BD, Petri WA Jr. Effect of substituting IPV for tOPV on immunity to poliovirus in Bangladeshi infants: An open-label randomized controlled trial. Vaccine. 2016 Jan 12;34(3):358-66. doi: 10.1016/j.vaccine.2015.11.046. Epub 2015 Nov 28. PMID 26643930
- [Result] Naylor C, Lu M, Haque R, Mondal D, Buonomo E, Nayak U, Mychaleckyj JC, Kirkpatrick B, Colgate R, Carmolli M, Dickson D, van der Klis F, Weldon W, Steven Oberste M; PROVIDE study teams; Ma JZ, Petri WA Jr. Environmental Enteropathy, Oral Vaccine Failure and Growth Faltering in Infants in Bangladesh. EBioMedicine. 2015 Sep 25;2(11):1759-66. doi: 10.1016/j.ebiom.2015.09.036. eCollection 2015 Nov. PMID 26870801
- [Derived] Ciszewski J, Taniuchi M, Lee B, Colgate ER, Platts-Mills JA, Haque R, Zaman K, Lopman B, Petri WA Jr, Kirkpatrick BD, Rogawski McQuade ET. Differences in Rotavirus Shedding and Duration by Infant Oral Rotavirus Vaccination Status in Dhaka, Bangladesh, 2011-2014. J Infect Dis. 2024 Jul 25;230(1):e75-e79. doi: 10.1093/infdis/jiad502. PMID 39052701
- [Derived] Kupkova K, Shetty SJ, Haque R, Petri WA Jr, Auble DT. Histone H3 lysine 27 acetylation profile undergoes two global shifts in undernourished children and suggests altered one-carbon metabolism. Clin Epigenetics. 2021 Sep 26;13(1):182. doi: 10.1186/s13148-021-01173-8. PMID 34565452
- [Derived] Lin Y, Zhou J, Kumar S, Xie W, G Jensen SK, Haque R, Nelson CA, Petri WA Jr, Ma JZ. Group penalized generalized estimating equation for correlated event-related potentials and biomarker selection. BMC Med Res Methodol. 2020 Aug 31;20(1):221. doi: 10.1186/s12874-020-01103-x. PMID 32867719
- [Derived] Williams FB, Kader A, Colgate ER, Dickson DM, Carmolli M, Uddin MI, Sharmin S, Islam S, Bhuiyan TR, Alam M, Nayak U, Mychaleckyj JC, Petri WA, Haque R, Qadri F, Kirkpatrick BD, Lee B. Maternal Secretor Status Affects Oral Rotavirus Vaccine Response in Breastfed Infants in Bangladesh. J Infect Dis. 2021 Oct 13;224(7):1147-1151. doi: 10.1093/infdis/jiaa101. PMID 32157282
- [Derived] Rogawski ET, Platts-Mills JA, Colgate ER, Haque R, Zaman K, Petri WA, Kirkpatrick BD. Quantifying the Impact of Natural Immunity on Rotavirus Vaccine Efficacy Estimates: A Clinical Trial in Dhaka, Bangladesh (PROVIDE) and a Simulation Study. J Infect Dis. 2018 Mar 5;217(6):861-868. doi: 10.1093/infdis/jix668. PMID 29514306
- [Derived] Lee B, Carmolli M, Dickson DM, Colgate ER, Diehl SA, Uddin MI, Islam S, Hossain M, Rafique TA, Bhuiyan TR, Alam M, Nayak U, Mychaleckyj JC, McNeal MM, Petri WA, Qadri F, Haque R, Kirkpatrick BD. Rotavirus-Specific Immunoglobulin A Responses Are Impaired and Serve as a Suboptimal Correlate of Protection Among Infants in Bangladesh. Clin Infect Dis. 2018 Jul 2;67(2):186-192. doi: 10.1093/cid/ciy076. PMID 29394355
- [Derived] Lee B, Dickson DM, deCamp AC, Ross Colgate E, Diehl SA, Uddin MI, Sharmin S, Islam S, Bhuiyan TR, Alam M, Nayak U, Mychaleckyj JC, Taniuchi M, Petri WA Jr, Haque R, Qadri F, Kirkpatrick BD. Histo-Blood Group Antigen Phenotype Determines Susceptibility to Genotype-Specific Rotavirus Infections and Impacts Measures of Rotavirus Vaccine Efficacy. J Infect Dis. 2018 Apr 11;217(9):1399-1407. doi: 10.1093/infdis/jiy054. PMID 29390150
- [Derived] Upfill-Brown A, Taniuchi M, Platts-Mills JA, Kirkpatrick B, Burgess SL, Oberste MS, Weldon W, Houpt E, Haque R, Zaman K, Petri WA Jr. Nonspecific Effects of Oral Polio Vaccine on Diarrheal Burden and Etiology Among Bangladeshi Infants. Clin Infect Dis. 2017 Aug 1;65(3):414-419. doi: 10.1093/cid/cix354. PMID 28444240
- [Derived] Lu M, Zhou J, Naylor C, Kirkpatrick BD, Haque R, Petri WA Jr, Ma JZ. Application of penalized linear regression methods to the selection of environmental enteropathy biomarkers. Biomark Res. 2017 Mar 9;5:9. doi: 10.1186/s40364-017-0089-4. eCollection 2017. PMID 28293424
- [Derived] Taniuchi M, Platts-Mills JA, Begum S, Uddin MJ, Sobuz SU, Liu J, Kirkpatrick BD, Colgate ER, Carmolli MP, Dickson DM, Nayak U, Haque R, Petri WA Jr, Houpt ER. Impact of enterovirus and other enteric pathogens on oral polio and rotavirus vaccine performance in Bangladeshi infants. Vaccine. 2016 Jun 8;34(27):3068-3075. doi: 10.1016/j.vaccine.2016.04.080. Epub 2016 May 3. PMID 27154394

RESULTS

PARTICIPANT FLOW:
Groups:
- Rotarix + IPV (Inactivated Polio Vaccine): Rotarix vaccine at 10 and 17 weeks of age plus IPV (inactivated polio vaccine) boost at 39 weeks in place of routine oral polio vaccine dose
- Rotarix + No IPV (Inactivated Polio Vaccine): Rotarix vaccine at 10 and 17 weeks of age and routine oral polio vaccine series
- No Rotarix + IPV (Inactivated Polio Vaccine): IPV (inactivated polio vaccine) boost at 39 weeks in place of routine oral polio vaccine dose
- No Rotarix + No IPV (Inactivated Polio Vaccine): No Rotarix vaccine and routine oral polio vaccine series
Period: Overall Study
Arm/Group | Rotarix + IPV (Inactivated Polio Vaccine) | Rotarix + No IPV (Inactivated Polio Vaccine) | No Rotarix + IPV (Inactivated Polio Vaccine) | No Rotarix + No IPV (Inactivated Polio Vaccine)
Started | 175 | 175 | 175 | 175
Completed | 153 | 150 | 141 | 151
Not Completed | 22 | 25 | 34 | 24
Not completed — Lost to Follow-up | 3 | 3 | 7 | 10
Not completed — Death | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 17 | 20 | 26 | 14
Not completed — Physician Decision | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Rotarix + IPV (Inactivated Polio Vaccine): Rotarix vaccine at 10 and 17 weeks of age plus IPV (inactivated polio vaccine) boost in place of the routine oral polio vaccine dose at 39 weeks
- Rotarix + No IPV (Inactivated Polio Vaccine): Oral Rotarix vaccine at 10 and 17 weeks of age and regular routine oral polio vaccine series
- No Rotarix + IPV (Inactivated Polio Vaccine): No Rotarix vaccine and IPV (inactivated polio vaccine) boost in place of the routine oral polio vaccine dose at 39 weeks
- Total: Total of all reporting groups
Arm/Group | Rotarix + IPV (Inactivated Polio Vaccine) | Rotarix + No IPV (Inactivated Polio Vaccine) | No Rotarix + IPV (Inactivated Polio Vaccine) | No Rotarix + No IPV (Inactivated Polio Vaccine) | Total
Number analyzed (Participants) | 175 | 175 | 175 | 175 | 700
Age, Continuous [Median (Full Range); unit: days] | 5 [1 to 7] | 5 [1 to 7] | 6 [1 to 7] | 5 [1 to 7] | 5 [1 to 7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 83 | 91 | 73 | 332
  Male | 90 | 92 | 84 | 102 | 368
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 175 | 175 | 175 | 175 | 700
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 175 | 175 | 175 | 175 | 700
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bangladesh | 175 | 175 | 175 | 175 | 700

OUTCOME MEASURES:

1. Primary Outcome: Presence of Fecal Shedding of Polio Vaccine Virus Determined by Culture (Polio Trial)
Description: Any Sabin type poliovirus in any fecal samples at days 0, 4, 11, 18 or 25 following week 52 dose
Time Frame: 25 days following week 52 visit
Population: Intention to treat. All participants analyzed as randomized
Measure: Count of Participants; unit: Participants
Groups:
- IPV (Inactivated Polio Vaccine): All who were randomized to receive IPV (inactivated polio vaccine) boost, regardless of whether they received Rotarix
- No IPV (Inactivated Polio Vaccine): All who were randomized to receive oral polio series only and no IPV (inactivated polio vaccine) boost dose, regardless of whether they received Rotarix
Arm/Group | IPV (Inactivated Polio Vaccine) | No IPV (Inactivated Polio Vaccine)
Number analyzed (Participants) | 350 | 350
Participants | 99 | 109
Statistical Analysis 1: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Test type: Superiority; p = 0.4, Chi-squared; 2 sided, not adjusted; Risk Difference (RD) = -2.9, 95% CI 2-sided [-9.6 to 3.9]

2. Primary Outcome: Number of Participants With One or More Episodes of Rotavirus-associated Diarrhea (Rotavirus Trial)
Description: Diarrheal episode defined as presence of 3 or more abnormally loose stools in 24h period with >=72 hours separating episodes. Rotavirus antigen detected by ELISA in diarrheal stool.
Time Frame: Birth to one year
Population: Intention to treat. All randomized participants are analyzed in the arms to which they were randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Rotarix: 2 dose oral Rotarix vaccine at week 10 and 17 regardless of whether IPV (inactivated polio vaccine) boost or not
- No Rotarix: No Rotarix vaccine, regardless of whether IPV (inactivated polio vaccine) boost or not
Arm/Group | Rotarix | No Rotarix
Number analyzed (Participants) | 350 | 350
Participants | 67 | 114
Statistical Analysis 1: Comparison: Rotarix vs No Rotarix; Test type: Superiority; p = 0.00004, Chi-squared — 2-sided, no adjustment; Risk Difference (RD) = 13.4, 95% CI 2-sided [7.0 to 19.8]

3. Secondary Outcome: Duration of Fecal Shedding of Polio Vaccine Virus, Each Sabin Type (Polio Trial)
Description: Shedding index, calculated as duration days multiplied by mean log (shedding amount) for Sabin types 1, 2, and 3.
  Outcome is conditioned on infants with at least one detection by quantitative PCR (qPCR) at day 4,11,18, or 25. If shedding data point was missing it was assumed that the infant was not shedding at that time.
  Lower shedding index is better outcome
Time Frame: from day 4 to day 25 following the week 52 visit
Population: This differs from the total population because it is a subset of total participants, limited to only those who shed the virus as determined by quantitative PCR assay (qPCR) Number analyzed differs from the number of participants shedding in outcome 5 (Presence of fecal polio virus shedding) because this shedding subset is determined using a different assay and time frame
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IPV (Inactivated Polio Vaccine): All who were randomized to receive IPV (inactivated polio vaccine) boost dose, regardless of whether they received Rotarix
Arm/Group | IPV (Inactivated Polio Vaccine) | No IPV (Inactivated Polio Vaccine)
Number analyzed (Participants) | 90 | 81
units on a scale
  Sabin type 1 | 17.9 (4.8) | 18.5 (4.5)
  Sabin type 2: number analyzed (Participants) | 63 | 49
  Sabin type 2 | 18.4 (4.7) | 19.6 (3.8)
  Sabin type 3: number analyzed (Participants) | 63 | 66
  Sabin type 3 | 17.7 (4.5) | 16.4 (4.4)
Statistical Analysis 1: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Sabin type 1 shedding; Test type: Superiority; p = 0.5, t-test, 2 sided; Mean Difference (Final Values) = 0.6
Statistical Analysis 2: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Sabin type 2 shedding; Test type: Superiority; p = 0.2, t-test, 2 sided; Mean Difference (Final Values) = 1.2
Statistical Analysis 3: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Sabin type 3 shedding; Test type: Superiority; p = 0.1, t-test, 2 sided; Mean Difference (Final Values) = -1.3

4. Secondary Outcome: Community Fecal Shedding of Polio Vaccine Virus Just Prior to Oral Polio Vaccine Dose at 52 Weeks (Polio Trial)
Description: Only 8 infants were shedding at baseline so results are not presented for this outcome due to insufficient data
Time Frame: post 52 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Presence of Fecal Polio Virus Shedding Within the Three Sabin Strains (Polio Trial)
Description: Frequency (%) of infants excreting poliovirus at any of the 5 time points (day 0, 4,11,18, 25) post week 52 oral polio vaccine dose.
  Presence of poliovirus is determined by polymerase chain reaction (PCR)
Time Frame: 25 days following week 52 visit
Population: Total Intention to treat population, all participants are included as randomized Number shedding differs from the number analyzed in outcome 3 (Duration of fecal shedding of polio vaccine virus) because shedding detection here is based on positive/negative PCR assay result
Measure: Count of Participants; unit: Participants
Arm/Group | IPV (Inactivated Polio Vaccine) | No IPV (Inactivated Polio Vaccine)
Number analyzed (Participants) | 350 | 350
Participants
  Sabin type 1 | 67 | 72
  Sabin type 2 | 22 | 33
  Sabin type 3 | 40 | 35
Statistical Analysis 1: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Sabin type 1; Test type: Superiority; Risk Difference (RD) = -1.4, 95% CI 2-sided [-7.3 to 4.5]
Statistical Analysis 2: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Sabin type 2; Test type: Superiority; Risk Difference (RD) = -3.1, 95% CI 2-sided [-7.2 to 0.9]
Statistical Analysis 3: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Test type: Superiority; Risk Difference (RD) = 1.4, 95% CI 2-sided [-3.2 to 6.1]

6. Secondary Outcome: Serum Neutralizing Antibody Response (Polio Trial)
Description: Seropositive defined as antibodies present at ≥1:8 dilution, antibody titers <1:8 were seronegative.
  Non-seroconversions are those who did not seroconvert between week 18 (post oral polio vaccine dose 2) and week 40, adjusted for residual maternal antibody
Time Frame: 18-40 weeks
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | IPV (Inactivated Polio Vaccine) | No IPV (Inactivated Polio Vaccine)
Number analyzed (Participants) | 233 | 215
Participants
  Non-seroconversion Sabin type 1: number analyzed (Participants) | 218 | 209
  Non-seroconversion Sabin type 1 | 9 | 79
  Non-seroconversion Sabin type 2: number analyzed (Participants) | 200 | 215
  Non-seroconversion Sabin type 2 | 9 | 62
  Non-seroconversion Sabin type 3 | 13 | 110
Statistical Analysis 1: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Test type: Superiority; Risk Difference (RD) = -33.7, 95% CI 2-sided [-40.7 to -26.5]
Statistical Analysis 2: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Test type: Superiority; Risk Difference (RD) = -24.3, 95% CI 2-sided [-31.1 to -17.5]
Statistical Analysis 3: Comparison: IPV (Inactivated Polio Vaccine) vs No IPV (Inactivated Polio Vaccine); Test type: Superiority; Risk Difference (RD) = -45.6, 95% CI 2-sided [-52.6 to -38.0]

7. Secondary Outcome: Total Number of Diarrheal Episodes (Rotavirus Trial)
Description: A diarrheal episode is defined as the presence of 3 or more abnormally loose stools in a 24 hour period with at least 72 diarrhea-free hours separating distinct episodes
Time Frame: Birth to one year
Population: Intention to treat population, included as randomized
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | Rotarix | No Rotarix
Number analyzed (Participants) | 350 | 350
episodes | 3 [1 to 5] | 3 [1 to 5]
Statistical Analysis 1: Comparison: Rotarix vs No Rotarix; Test type: Superiority; p = 0.981, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Total Duration of Rotavirus-associated Diarrheal Episodes (Rotavirus Trial)
Description: A diarrheal episode is defined as the presence of 3 or more abnormally loose stools in a 24 hour period with at least 72 diarrhea-free hours separating distinct episodes.
  Rotavirus positive specimens were determined by ELISA Those with no rotavirus diarrheal episodes are counted as duration 0
Time Frame: Birth to one year
Population: Intention to treat, all included as randomized
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Rotarix | No Rotarix
Number analyzed (Participants) | 350 | 350
days | 0 [0 to 0] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Rotarix vs No Rotarix; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Birth to one year
Groups:
- Rotarix + IPV: Rotarix vaccine at 10 and 17 weeks of age plus inactivated polio vaccine in place of the routine oral polio vaccine dose at 39 weeks
- Rotarix + No IPV: Rotarix vaccine at 10 and 17 weeks of age and routine oral polio vaccine series
- No Rotarix + IPV: No Rotarix vaccine and inactivated polio vaccine in place of the routine oral polio vaccine dose at 39 weeks
- No Rotarix + No IPV: No Rotarix vaccine and routine oral polio vaccine series
Arm/Group | Rotarix + IPV | Rotarix + No IPV | No Rotarix + IPV | No Rotarix + No IPV
All-Cause Mortality (participants affected / at risk) | 2/175 | 2/175 | 1/175 | 0/175
Serious Adverse Events (participants affected / at risk) | 16/175 | 16/175 | 20/175 | 21/175
Other Adverse Events (participants affected / at risk) | 0/175 | 0/175 | 0/175 | 0/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rotarix + IPV (N=175) | Rotarix + No IPV (N=175) | No Rotarix + IPV (N=175) | No Rotarix + No IPV (N=175)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 14 (15) | 17 (17) | 17 (19)
Respiratory illness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile Illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Inguinal heria (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Convulsions (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No